CLINICAL TRIAL: NCT05325697
Title: Combining Oral Nutrition Supplementation With a Multicomponent Exercise Program in Elderly Malnourished Frail Patients After Hospital Stay A Feasibility Study
Brief Title: Combining Nutrition Supplementation With an Exercise Program in Elderly Malnourished Frail Patients After Hospital Stay
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Department of Geriatric Medicine FELIX PLATTER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-01058
Record Dates: First submitted 2022-02-23; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Frailty; Sarcopenia; Malnutrition; Protein
Keywords: Elderly; Exercise program; Oral Nutrition Supplementation
MeSH Terms: conditions — Frailty; Sarcopenia; Kwashiorkor

STUDY DESIGN:
Intervention Model Description: Single-arm, open label feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single - Arm (Experimental): 12 weeks intervention with a combined physical exercise program (vivifrail) and oral nutritional supplementation (Moltein Plus)
  Interventions: Combination Product: Intervention consisting of a multicomponent exercise program combined with an oral nutritional supplement

INTERVENTIONS:
Combination Product: Intervention consisting of a multicomponent exercise program combined with an oral nutritional supplement — The multicomponent exercise program to prevent frailty and risk of falls (Vivifrail) was developed by a European expert group co-funded by the ERASMUS+ programm of the European Union. The program consists of a screening and a subsequent 12-week exercise program. The screening classifies individuals into four categories: disabled, frail, pre-frail, or robust and the difficulty of the program's exercises is adapted to the categories and it includes endurance, balance, and resistance training as well as stretching exercises. This exercise program will be combined with an oral nutritional supplement (Moltein®Plus), which was specifically designed to promote muscle health in elderly people. Moltein®Plus is completely balanced oral nutrition supplement made from whey protein fortified with leucine. Enriching dietary protein with leucine allows to maximize muscle protein synthesis rates without calling for very high protein doses, which are difficult to ingest for older individuals.

SUMMARY:
The objective of this study is to investigate the feasibility of a combined nutritional and home-based exercise intervention in elderly, malnourished, frail patients after hospital discharge.

Adherence to exercise program, adherence to oral nutrition supplement, potential inhibiting factors to follow exercise program, changes in nutritional status, muscle mass and function, quality of life are outcome factors.

The intervention consists of 12 weeks with a physical exercise program (vivifrail) and oral nutritional supplementation (Moltein Plus).

The investigators hypothesize that 12 weeks of a combined nutritional and home-based multicomponent exercise program is feasible for frail elderly patients after hospital discharge, meaning that ≥70% of the exercise sessions will be completed and oral supplements will be consumed by the participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65
* Malnutrition: Nutrition Risk Screening ≥3
* Frail/pre-frail status according Fried Frailty Phenotype: 1-2 criteria present = pre frail, > 2 criteria present = frail
* Frailty status according to SPPB: A: 0-3 points = disabled, B (B+): 4-6 points = frail (at risk of falls), C (C+): 7-10 points = pre-frail (at risk of falls), D: 10-12 points = robust.
* Ability to sit
* Consent to participate in the study
* Ability to follow the instructions of the vivifrail program
* Prescription for use of an ONS

Exclusion Criteria:

* Severe acute cardiovascular issues: eg. unstable angina pectoris, uncontrolled arrhythmia, uncontrolled arterial hypertension or unstable cardiovascular disease or other unstable medical condition.
* Persisting oedema and/or ascites
* Contraindication for the protein-rich ONS (e.g. cow's milk allergy, end stage renal disease without renal replacement therapy) or dysphagia for liquids
* non-removable plasters or bandages at feet or hands aggravating body impedance analysis (BIA), implanted defibrillation device
* Parenteral/tube feeding
* No access to telephone or severe hearing loss
* Terminal illness
* Hospitalized due to pulmonary thromboembolism
* Considerable cognitive impairment: Mini-mental score < 18 or advice of healthcare professionals against inclusion due to cognitive or psychological reasons.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to the combined exercise program with the oral nutrition supplement: Self-admistered questionnaire | The questionnaire is completed daily from the first day after hospital discharge until the last day of the 12-week intervention (84 days).
  Subjects will use a self-admistered questionnaire in paper pencil form consisting of the combined vivifrail passport checklist (provided by the vivifrail program, asking if the exersise program was performed or not and a 3-point likert scale question: "How demanding were the exercises for you?" with the answer options very demanding, moderately demanding and not very demanding) and a oral nutrition checklist (asking if the oral supplementation was consumed or not) to keep record of completed exercise sessions as well as the effort perceived during the activities and the daily intake of the oral nutritional supplementation. Higher scores of absolved exercise sessions with the intake of the oral nutrition mean a better outcome.
Inhibiting factors to follow the combined exercise and nutritional program: Semi-structured phone call interview using a self developed questionnaire | 1 week after the initiation of the program (first day after hospital discharge plus 7 days)
  The semi-structured phone interviews have the purpose to shed light on the difficulties participants encountered while following the intervention. The self developed questionnaire (adapted from Hoogland J et al. 2019) uses a semi-structured approach and consists of 10 questions: Have you forgotten to consume ONS in the last 7 days? What is the usual dose per day you have taken in the last 7 days? When do you consume the drinkable food? How and when do you usually consume the ONS? Have you forgotten to exercise in the last 7 days? Did you complete the entire exercise session, or did you skip some exercises? What were the reasons that made it difficult to start or finish an exercise session in the last 7 days? How many minutes did it take to do the exercises per day? Do you feel stronger now than before you started the exercise and nutrition program? Do you feel less likely to fall now than before you started the exercise and nutrition program?
Inhibiting factors to follow the combined exercise and nutritional program: Semi-structured phone call interview using a self developed questionnaire | 4 weeks after the initiation of the program (first day after hospital discharge plus 28 days)
  The semi-structured phone interviews have the purpose to shed light on the difficulties participants encountered while following the intervention. The self developed questionnaire (adapted from Hoogland J et al. 2019) uses a semi-structured approach and consists of 10 questions: Have you forgotten to consume ONS in the last 7 days? What is the usual dose per day you have taken in the last 7 days? When do you consume the drinkable food? How and when do you usually consume the ONS? Have you forgotten to exercise in the last 7 days? Did you complete the entire exercise session, or did you skip some exercises? What were the reasons that made it difficult to start or finish an exercise session in the last 7 days? How many minutes did it take to do the exercises per day? Do you feel stronger now than before you started the exercise and nutrition program? Do you feel less likely to fall now than before you started the exercise and nutrition program?
Inhibiting factors to follow the combined exercise and nutritional program: Semi-structured phone call interview using a self developed questionnaire | 8 weeks after the initiation of the program (first day after hospital discharge plus 56 days)
  The semi-structured phone interviews have the purpose to shed light on the difficulties participants encountered while following the intervention. The self developed questionnaire (adapted from Hoogland J et al. 2019) uses a semi-structured approach and consists of 10 questions: Have you forgotten to consume ONS in the last 7 days? What is the usual dose per day you have taken in the last 7 days? When do you consume the drinkable food? How and when do you usually consume the ONS? Have you forgotten to exercise in the last 7 days? Did you complete the entire exercise session, or did you skip some exercises? What were the reasons that made it difficult to start or finish an exercise session in the last 7 days? How many minutes did it take to do the exercises per day? Do you feel stronger now than before you started the exercise and nutrition program? Do you feel less likely to fall now than before you started the exercise and nutrition program?
Inhibiting factors to follow the combined exercise and nutritional program: Semi-structured phone call interview using a self developed questionnaire | 12 weeks after the initiation of the program (first day after hospital discharge plus 84 days)
  The semi-structured phone interviews have the purpose to shed light on the difficulties participants encountered while following the intervention. The self developed questionnaire (adapted from Hoogland J et al. 2019) uses a semi-structured approach and consists of 10 questions: Have you forgotten to consume ONS in the last 7 days? What is the usual dose per day you have taken in the last 7 days? When do you consume the drinkable food? How and when do you usually consume the ONS? Have you forgotten to exercise in the last 7 days? Did you complete the entire exercise session, or did you skip some exercises? What were the reasons that made it difficult to start or finish an exercise session in the last 7 days? How many minutes did it take to do the exercises per day? Do you feel stronger now than before you started the exercise and nutrition program? Do you feel less likely to fall now than before you started the exercise and nutrition program?

SECONDARY OUTCOMES:
Changes in nutritional status using the MNA-LF | The MNA-LF is measured at baseline, within one week before hospital discharge
  Changes in nutritional status will be measured using the MNA-LF(Mini Nutritional Assessment Long Format).
  The MNA-LF scale ranges from 0-30 points: 24-30 points: normal status, 17-23.5 points: risk for malnutrition, <10 points: malnutrition.
Changes in nutritional status using the MNA-LF | The MNA-LF is measured 12 weeks (84days) after the initiation of the intervention
  Changes in nutritional status will be measured using the MNA-LF(Mini Nutritional Assessment Long Format).
  The MNA-LF scale ranges from 0-30 points: 24-30 points: normal status, 17-23.5 points: risk for malnutrition, <10 points: malnutrition.
Muscle mass | The BIA at baseline is performed within one week before hospital discharge
  For evaluation of muscle mass, Bioelectrical impedance analysis (BIA) is performed in all included patients using a BIVA 101® (Akern, SMT medical GmbH, Würzburg, Germany). It measures the apendicular muscle mass. The cut-off values for sarcopenia are: ♂< 20 kg, 7 kg/m2, ♀ < 16 kg, 5.5 kg/m2.
Muscle mass | The BIA is measured 12 weeks (84days) after the initiation of the intervention
  For evaluation of muscle mass, Bioelectrical impedance analysis (BIA) is performed in all included patients using a BIVA 101® (Akern, SMT medical GmbH, Würzburg, Germany). It measures the apendicular muscle mass. The cut-off values for sarcopenia are: ♂< 20 kg, 7 kg/m2, ♀ < 16 kg, 5.5 kg/m2.
EQ-5D-3L Quality of life | Quality of life is measured within one week before hospital discharge
  Quality of life will be measured with the EQ-5D-3L questionnaire intepreted according to the EuroQol guidelines.
EQ-5D-3L Quality of life | Quality of life is measured 12 weeks (84days) after the initiation of the intervention
  Quality of life will be measured with the EQ-5D-3L questionnaire intepreted according to the EuroQol guidelines.
Frailty assessment | SPPB is measured within one week before hospital discharge
  The Short Physical Performance Battery (SPPB) is a group of measures that combines the results. of the gait speed, chair stand and 3 balance tests (Guralnik et al., 2000). It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. Scores range from 0 to 12 points, ≤ 9 points indicate physical frailty, ≤ 8 points indicate severe sarcopenia, ≤ 3 points indicate severe limitations in the activities of daily living.
Frailty assessment | SPPB is measured 12 weeks (84days) after the initiation of the intervention
  The Short Physical Performance Battery (SPPB) is a group of measures that combines the results. of the gait speed, chair stand and 3 balance tests (Guralnik et al., 2000). It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. Scores range from 0 to 12 points, ≤ 9 points indicate physical frailty, ≤ 8 points indicate severe sarcopenia, ≤ 3 points indicate severe limitations in the activities of daily living.
Hand grip strenght | Hand grip strength is measured within one week before hospital discharge
  Hand grip strength is assessed using a Martin Vigorimeter. The Martin Vigorimeter is a pseudodynamic dynamometer that measures the pressure when subjects press a rubber bulb connected by a tube to a manometer, with pressure being expressed in kiloPascal (kPa). Higher scores mean a better outcome. Cut-off points for poor muscle strength in the assessment for sarcopenia are: female 27 kPa, male 45 kPa.
Hand grip strenght | Hand grip strength is measured 12 weeks (84days) after the initiation of the intervention
  Hand grip strength is assessed using a Martin Vigorimeter. The Martin Vigorimeter is a pseudodynamic dynamometer that measures the pressure when subjects press a rubber bulb connected by a tube to a manometer, with pressure being expressed in kiloPascal (kPa). Higher scores mean a better outcome. Cut-off points for poor muscle strength in the assessment for sarcopenia are: female 27 kPa, male 45 kPa.
Timed up and go assessment to assess functional ability and mobility | TUG is assessed within one week before hospital discharge
  The timed up and go (TUG) assessment assesses functional ability and mobility. The probands start the assessment in a seated position, then stand up upon the assessor's command, walk 3 meters, turn around, walk back to the chair and sit down. Time measurement (seconds) starts when the back of the participant leaves the backrest and is stopped when is back seated. An older adult who takes ≥12 seconds to complete the TUG is at risk for falling. Lower scores indicate better outcomes. ≥20 seconds to complete the TUG indicate severe sarcopenia.
Timed up and go assessment to assess functional ability and mobility | TUG is assessed 12 weeks (84days) after the initiation of the intervention
  The timed up and go (TUG) assessment assesses functional ability and mobility. The probands start the assessment in a seated position, then stand up upon the assessor's command, walk 3 meters, turn around, walk back to the chair and sit down. Time measurement (seconds) starts when the back of the participant leaves the backrest and is stopped when is back seated. An older adult who takes ≥12 seconds to complete the TUG is at risk for falling. Lower scores indicate better outcomes. ≥20 seconds to complete the TUG indicate severe sarcopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Reto W Kressig, Prof., Principal Investigator — University Department of Geriatric Medicine

IPD SHARING:
Plan to Share IPD: No